CLINICAL TRIAL: NCT06769815
Title: Host Immunity, Plasmodium and Pathogens Co-Infections
Acronym: HIPPI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut de Recherche pour le Developpement (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-079; IRB2024-01 (Other: IRB00006966 Institut Pasteur IRB #1); 043/2024/CBRS (Other: Comité de Bioéthique pour la Recherche en Santé)
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Malaria; Bacterial Co-infection
Keywords: malaria; co-infection; immune response; epigenetic mechanisms; children; Togo
MeSH Terms: conditions — Malaria; Coinfection | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Febrile and non febrile children, pregnant women and new borns (Other): The study population is composed of children under the age of 5, which is also the population most at risk of malaria, living in the endemic areas of Lomé and Tsévié in Togo.
  Interventions: Other: Blood sample; Other: Urine sample; Other: oropharyngeal sample; Other: Optionnal : stool sample; Other: Optionnal : cerebrospinal fluid; Other: placental biopsy

INTERVENTIONS:
Other: Blood sample — For febrile children at the time of inclusion : 6.25 ml to 8.25 ml of blood ; For non febrile children at the time of inclusion : 4 ml of blood ; For pregnant women at the time of inclusion : 5 ml of peripheral blood, 5 ml of placental blood, 20 to 40 ml of umbilical cord blood ; For new borns : drop of blood on child's heel each month and 5 ml of blood the 12th and last month.
Other: Urine sample — For febrile children : 10 ml of urine
Other: oropharyngeal sample — For febrile children : oropharyngeal swab sampling
Other: Optionnal : stool sample — For febrile children (only as part of the care of the child) : 5g stool
Other: Optionnal : cerebrospinal fluid — For febrile children (only as part of the care of the child in case of suspected meningitis) : 4 additional drops of cerebrospinal fluid
Other: placental biopsy — For pregnant women : placental biopsy the size of 2 rice grains

SUMMARY:
Few studies have focused on malaria co-infections, mainly caused by Plasmodium falciparum, occurring mainly in children under 5 years of age in sub-Saharan Africa. These studies have focused on malaria-associated bacterial sepsis, with an estimated prevalence of 9.1% and associated mortality of 15.0%. However, no study has documented infectious sites other than the blood compartment, considered viruses and parasites as possible causes of infection in addition to bacteria, and used molecular diagnostic methods based on PCRs, which are more sensitive. Thus, the prevalence of these co-infections and the spectrum of pathogens involved are probably underestimated, as is the impact of these co-infections on mortality. Furthermore, it has been shown that malaria infections can condition the immune cells of naturally exposed individuals, potentially leading to greater susceptibility to all types of infection. But these mechanisms have never been documented in the context of co-infections.

The WHO recommends the use of broad-spectrum antibiotics in cases of severe malaria, in addition to antimalarial drugs, as it can be difficult to differentiate clinically between severe malaria and severe bacterial infection (bacteremia, pneumonia and meningitis). Yet this empirical use of antibiotics could be contributing to an increase in antibiotic resistance. Identifying the determinants of co-infection with malaria and severe bacterial infection would enable this treatment to be better targeted.

These determinants remain undetermined as no study has considered other causes of severe bacterial infection other than bacteremia, used appropriate statistical methodology (univariate analysis only) and explored important determinants, notably the capacity of children's innate immunity to respond to severe bacterial infection.

DETAILED DESCRIPTION:
This is a prospective multicenter longitudinal study.

The study will focus on several populations:

* febrile children: aged between 6 and 60 months consulting ;
* non-febrile children: aged between 6 and 60 months consulting.
* Pregnant women.
* newborns: those born to mothers included in the study with or without pregnancy-associated malaria.

The study will be based on :

* Clinical and microbiological documentation of acute febrile episodes in recruited children
* Documentation of vital status in children 3 months after recruitment
* Ability of host cells to respond to infections.

ELIGIBILITY:
Inclusion Criteria:

Febrile children:

* aged between 6 and 60 months
* with a febrile episode lasting less than 7 days (axillary temperature >=37.5° Celsius)
* whose state of health is compatible with a minimum single blood sample volume of 6.25 ml

Non-febrile children:

* aged between 6 and 60 months
* with axillary temperature <37.5° Celsius
* no clinical signs of infection at the time of inclusion
* no infectious episode or fever for 7 days

Pregnant women :

* giving birth in the project's partner health center
* intending to reside in the study area during the newborn follow-up period
* with a mono-fetal pregnancy
* With an apparently uncomplicated delivery not requiring referral to a higher-level health facility

Newborns at delivery:

* Born at term (determined by Ballard score)
* whose parents or legal guardians reside in the study area during the newborn's follow-up period

Exclusion Criteria:

For all :

- person already participating in another biomedical research project.

For febrile and non-febrile children:

- chronic non-infectious pathology (cancer, malnutrition, etc.)

For pregnant women

* scheduled caesarean section for current pregnancy
* Caesarean section in previous pregnancies
* chronic non-infectious pathology during pregnancy (diabetes, hypertension, pre-eclampsia)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Determine the extent and microbiological spectrum of malaria co-infections in children under 5. | 3 years
  the number of malaria co-infection events in febrile children.

SECONDARY OUTCOMES:
Assess the impact of malaria co-infections on mortality | 2 years
  Number of deaths in children under 5 with malaria co-infection
Identify the underlying immunological mechanisms mediating malaria co-infections | 2 years
  Concentration of cytokines IL6, IL1β and TNFα and IL 10 in children under 5 years of age
Identify epigenetic and transcriptomic modifications in infant, maternal and placental blood cells mediating malaria co-infections | 2 years
  Expression level of transcripts according to the populations studied will be measured by RNA-seq
Identify molecules associated with epigenetic modifications (metabolome, proteome). | 2 years
  Expression level of proteins and metabolites according to the populations studied will be measured by RNA-seq
Identify determinants of malaria co-infections and severe bacterial infections. | 2 years
  The number of malaria co-infection events associated with severe bacterial infection in febrile children under 5 years of age.

CONTACTS AND LOCATIONS:
Overall Officials: Bich-Tram Huynh, PhD, Study Director — Institut Pasteur; Luc Douti, MD, Principal Investigator — CHU-Campus de Lomé; Serge Ekoué Gbadoe, MD, Principal Investigator — Hôpital de district Polyclinique de Zio-Tsévié